# STUDY PROTOCOL WITH STATISTICAL ANALYSIS PLAN

**Study Title:** Vaginal Breech Birth Management: serious mobile game design and evaluation for midwifery students

NCT Number: NCT05551611

**Document Date:** March 14, 2025

1. Background and Rationale

Vaginal breech birth (VBB) is now an infrequent clinical event; consequently, midwifery

students have limited real-life learning opportunities. Serious games offer cost-effective,

repeatable simulation experiences that can enhance knowledge acquisition. This study evaluates

a bespoke mobile serious game designed to teach VBB management and compares it with

traditional lecture-based instruction.

2. Aims

• To determine whether the serious mobile game improves short-term knowledge of VBB

management compared with a traditional lecture.

To compare knowledge retention at 14 days and 7 months post-intervention between

groups.

3. Study Design

Prospective, parallel-group, randomised controlled quasi-experimental trial with

pre-test/post-test assessments.

• Setting: Midwifery departments of two Turkish universities (Kocaeli University &

Eskişehir Osmangazi University).

**Duration**: February 2022 – December 2022 (follow-up to July 2023).

4. Study Population and Eligibility Criteria

Third-year midwifery students.

Inclusion:

Completed "Normal Childbirth & Postpartum" course.

Provide written informed consent.

**Exclusion**: Previous theoretical or practical training on breech presentation.

5. Interventions

5.1. Experimental Arm – "Game Group"

Students play the Vaginal Breech Birth Management Serious Mobile Game once ( $\approx 30$ –45 min) under supervised classroom conditions. Headphones supplied; individual play; no time limit.

## 5.2. Control Arm – "Lecture Group"

Traditional 45-min lecture covering identical VBB content, delivered by the same investigator with slides & discussion.

#### 6. Outcome Measures

| Type | Name | Description | Scale (range) | Direction |
|---|---|---|---|---|
| Primary | Vaginal Breech Birth Management Knowledge Test | 47-item multiple-choice test assessing knowledge of trauma & management in VBB. Each correct answer = 1 point; Total score 0–47. No subscales; higher scores = better knowledge/outcome. | 0–47 scores<br>on a scale | Higher = better |

Assessments at baseline (pre-test), Day 0 (immediately after intervention), Day 14, and Month 7.

## 7. Sample Size & Power Calculation

Using Day 0 pilot means (Game= $40.5\pm4.2$ ; Control= $37.8\pm5.1$ ),  $\alpha=0.05$ , two-sided Mann–Whitney U, power=0.80 required **n=35 per group**. Allowing 10 % attrition, recruitment target set at 40 per group (total 80). Final analysed: Game=39; Control=40.

#### 8. Randomisation and Allocation

Simple randomisation (1:1) using computer-generated list by independent statistician. Group assignment placed in sealed opaque envelopes; opened by researcher immediately before session.

### 9. Data Collection Procedures

Knowledge test administered on paper. Unique codes used instead of names. Data entered twice into SPSS 20.0; discrepancies resolved by audit.

## 10. Statistical Analysis Plan (SAP)

#### 10.1. Primary Outcome Analysis

- **Between-group comparison (Day 0)**: Mann–Whitney U test.
- Report Median (IQR) & Mean  $\pm$  SD.

## 10.2. Secondary/Exploratory Analyses

- Within-group change over time: Friedman two-way repeated measures ANOVA (pre, Day 0, Day 14, Month 7). Post-hoc Dunn-Bonferroni pairwise tests.
- Between-group at Day 14 & Month 7: Mann-Whitney U.

## 10.3. Assumptions & Checking

• Normality checked via Shapiro–Wilk; non-normal distribution anticipated ⇒ non-parametric tests chosen.

#### 10.4. Handling Missing Data

Complete-case analysis. Participants with missing follow-up tests excluded from that specific time-point analysis; no imputation performed (anticipated < 5 % missing).

#### 10.5. Software

IBM SPSS Statistics v20.0 (Armonk, NY, USA).

## 10.6. Interim Analysis

None planned; single-session educational intervention with minimal risk.

#### 11. Ethical Considerations

Ethics approval: Kocaeli University Non-Interventional Clinical Research Ethics Committee (28 Jan 2022; GOKAEK-2022/02.11). Study conducted by Declaration of Helsinki. Written informed consent obtained. Data anonymised.

# 12. Data Monitoring & Safety

Minimal-risk educational study; no independent DSMB. Adverse events unlikely; any unanticipated problems to be reported to ethics committee within 7 days.

#### 13. Administrative Information & Protocol Amendments

All substantial amendments approved by ethics committee and recorded in ClinicalTrials.gov history.